CLINICAL TRIAL: NCT00930371
Title: Effect of Diet Composition on Liver Fat and Glucose Metabolism
Acronym: DietLFAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kristina Utzschneider, Associate Professor of Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 35016-D
Record Dates: First submitted 2009-06-26; First posted 2009-06-30 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Fatty Liver
Keywords: fatty liver; insulin resistance; diet; inflammation; oxidative stress
MeSH Terms: conditions — Fatty Liver; Insulin Resistance; Inflammation | interventions — Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: high fat/high saturated fat diet — 4 weeks 55% fat/25% saturated fat isocaloric diet
  Other Names: Diet
Other: low fat/low saturated fat diet — 4 weeks 20% fat/8% saturated fat isocaloric diet
  Other Names: Diet

SUMMARY:
This study is designed to determine if the amount of fat and saturated fat in the diet contributes to the development of a condition called fatty liver disease in the absence of changes in weight.

DETAILED DESCRIPTION:
A condition called non-alcoholic steatohepatitis is characterized by fat accumulation in the liver and associated inflammation. This condition is strongly associated with obesity, insulin resistance and type 2 diabetes. Diets high in saturated fat result in fatty liver, insulin resistance and liver injury in animal models. Dietary composition may contribute not only to hepatic fat accumulation and insulin resistance but may also promote inflammation leading to chronic liver disease in humans. This study will test the hypothesis that a diet high in fat and saturated fat contributes to liver fat accumulation, insulin resistance and inflammation by comparing the effects of a four-week, weight stable high fat/high saturated fat diet (55% calories from fat/25% saturated fat) with a four-week, weight stable low fat/low saturated fat diet (20% fat/8% saturated fat) in overweight and obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years old, men and women, otherwise in good general health, BMI >27 kg/m2

Exclusion Criteria:

* Abnormal glucose tolerance, fasting glucose>100 mg/dl or diabetes
* History of liver condition or alanine aminotransferase (ALT) above the upper limit of the normal range
* Use of medications that cause insulin resistance or fatty liver: niacin, glucocorticoids, estrogens, tamoxifen, amiodarone, accutane, sertraline, atypical antipsychotics, anti-HIV medications
* Chronic use of anti-inflammatory medications (aspirin, ibuprofen, naprosyn, steroids, etc)
* Average alcohol intake >20 grams/day
* Tobacco use
* Creatinine >1.5 mg/dl for men and >1.4 mg/dl for women
* Hematocrit <33%
* Pregnancy or lactation
* Significant weight loss within the past 6 months (>5% body weight)
* Claustrophobia or any contraindications to being placed in the magnet for the MRS scan such as pacemakers, defibrillators, brain aneurysm clips, etc.
* Other serious medical conditions or inflammatory conditions such as cancer, inflammatory arthritis, etc.
* History of multiple food allergies or intolerances or severe food allergies
* History of coronary artery disease, history of or treatment of hyperlipidemia, LDL >200 mg/dl, fasting triglycerides >300 mg/dl
* Weight >300 pounds

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
hepatic triglyceride content by MRS | 4 weeks

SECONDARY OUTCOMES:
insulin sensitivity | 4 weeks
systemic and subcutaneous adipose tissue inflammation | 4 weeks
oxidative stress markers | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kristina M Utzschneider, MD, Principal Investigator — VA Puget Sound Health Care System/University of Washington
Locations (2):
- United States (2):
  - University of Washington, Seattle, Washington
  - VA Puget Sound Health Care System, Seattle, Washington

REFERENCES:
- [Result] Marina A, von Frankenberg AD, Suvag S, Callahan HS, Kratz M, Richards TL, Utzschneider KM. Effects of dietary fat and saturated fat content on liver fat and markers of oxidative stress in overweight/obese men and women under weight-stable conditions. Nutrients. 2014 Oct 28;6(11):4678-90. doi: 10.3390/nu6114678. PMID 25353663
- [Result] von Frankenberg AD, Marina A, Song X, Callahan HS, Kratz M, Utzschneider KM. A high-fat, high-saturated fat diet decreases insulin sensitivity without changing intra-abdominal fat in weight-stable overweight and obese adults. Eur J Nutr. 2017 Feb;56(1):431-443. doi: 10.1007/s00394-015-1108-6. Epub 2015 Nov 28. PMID 26615402